CLINICAL TRIAL: NCT02082587
Title: Pilot Study of the Toronto Brief Neurocognitive Battery (BNB)
Brief Title: Toronto BNB Pilot Study
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: OCREB 14-006
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Brain Metastases
Keywords: brain metastases; brain mets; WBRT
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- QOL Assessment

SUMMARY:
As treatments improve and patients live longer with cancer, even after it has spread to the brain, efforts to improve quality of life are growing. Neurocognitive function (thinking ability and memory) is an area of particular concern for patients with brain metastases (cancer that can spread to the brain). Although there are established tests to measure neurocognitive function, these require a face-to-face assessment and can take a long time to complete. As a result, efforts to use these tests to measure changes in neurocognitive function in patients following treatment for brain metastases have resulted in a large proportion of patients who do not return for follow-up. This has limited the ability to evaluate the impact of current treatments on neurocognitive function. This study aims to evaluate a shorter, telephone-based neurocognitive assessment tool, which would make it easier for patients to complete these tests in follow-up. If this new tool is found to reliably measure neurocognitive function, it could be used for future studies evaluating new interventions that prevent or treat neurocognitive deterioration following treatment of brain metastases. This is the first prospective study to evaluate the feasibility and reliability of a novel telephone-based brief neurocognitive assessment battery (Toronto BNB) compared with the same battery delivered face-to-face in this population. The investigators hypothesize that telephone administration of this brief neurocognitive battery will reliably evaluate neurocognitive function and improve patient ability to complete follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years old) with newly diagnosed brain metastases planned for whole brain radiotherapy
* Performance status ECOG 0-2
* English-speaking (due to small sample-size in this pilot study, only English testing will be completed)

Exclusion Criteria:

* Prior whole brain radiotherapy
* Presence of any condition which can prevent completion of neurocognitive assessment, including:
* Hearing impairment which is sufficient to prevent the patient from comprehending English instructions in a quiet environment
* Major psychiatric diagnosis or neurological condition associated with cognitive impairment which, in the judgement of the investigator, would make the patient inappropriate for study participation (e.g., schizophrenia, multiple sclerosis, Parkinson's disease, prior ischemic stroke, dementia, traumatic brain injury with loss of consciousness for greater than 30 minutes, expressive/receptive aphasia, developmental delay)
* Patients with planned systemic therapy or additional radiotherapy within the interval between clinic and telephone Toronto BNB testing
* Minimal English skills such that subjects would be unable to follow simple English instructions (either verbal or written) or be unable to read questionnaires of a grade 8 standard with the help of a research assistant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed brain metastases planned for whole brain radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-09; Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Evaluate feasibility of utilizing a telephone assessment in patients with brain metastases | 1.5 years
  The telephone-based tool will be considered feasible if the proportion of participants who complete baseline and follow-up telephone-based assessments is the same as or greater than the proportion of participants who complete the in-clinic assessments.
Evaluate the interprocedure (telephone vs. clinic) reliability | 1.5 years
  Cronbach's alpha coefficient at each time point (baseline, 1 month, 4 months) will be calculated to assess the following z scores: Patient results from individual neurocognitive tests will be converted to a z score (the number of standard deviations above or below the mean). Overall averaged global z scores will be compared between the telephone and clinic assessments using the Toronto BNB. Cronbach's alpha coefficient will be evaluated as follows: 0-0.2 poor agreement; 0.3-0.4 fair agreement; 0.5-0.6 moderate agreement; 0.7-0.8 strong agreement; >0.8 very strong agreement.

SECONDARY OUTCOMES:
Evaluate the change in neurocognitive function before and after WBRT using the Toronto BNB | 1.5 years
  Paired t-tests will be used to assess whether any statistically significant change is observed between neurocognitive scores obtained at 1 month and 4 months after WBRT as compared to baseline (before WBRT)
Evaluate sensitivity to change (responsiveness) of the Toronto BNB (in clinic and by telephone) | 1.5 years
  Paired t-tests will be used to assess whether any statistically significant change is observed between 1 month and 4 months using the BNB obtained in clinic and then using the BNB obtained over the phone.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chung, MD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Sunnybrook Hospital - Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario